CLINICAL TRIAL: NCT03755752
Title: Safety of Trypan Blue Capsule Staining to Corneal Endothelium in Patients With Diabetic Retinopathy
Brief Title: Safety of Trypan Blue on Endothelium of Diabetic Retinopathy Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Khaled Abdelazeem, Lecturer of Ophthalmology, Assiut University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 17300250
Record Dates: First submitted 2018-11-26; First posted 2018-11-28 (Actual); Last update posted 2018-11-28 (Actual); Status verified 2018-11

CONDITIONS: Cataract Diabetic
MeSH Terms: interventions — Phacoemulsification; Trypan Blue; Staining and Labeling

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Randomization was done using an envelope technique wherein, after each patient was placed on the operating bed, the surgeon opened the patient's corresponding envelope, which contained information about whether Trypan Blue should be used for anterior capsular staining or not.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phacoemulsification with Trypan Blue (Experimental): Phacoemulsification with Trypan Blue capsule staining of the anterior lens capsule in patients with diabetic retinopathy
  Interventions: Procedure: Phacoemulsification with and without Trypan Blue capsule staining
- Phacoemulsification without Trypan Blue (Experimental): Phacoemulsification without Trypan Blue capsule staining of the anterior lens capsule in patients with
  Interventions: Procedure: Phacoemulsification with and without Trypan Blue capsule staining

INTERVENTIONS:
Procedure: Phacoemulsification with and without Trypan Blue capsule staining — Phacoemulsification for patients with diabetic retinopathy having cataract in both eyes. One eye underwent phacoemulsification with trypan blue capsule staining and the other eye underwent phacoemulsification without trypan blue.

SUMMARY:
This study examines the use of Trypan Blue staining of the corneal endothelium in patients undergoing phacoemulsification. It is a single-center prospective, randomized individual cohort study. One eye in each patient with diabetic retinopathy will undergo phacoemulsification without Trypan Blue capsule staining (control eye) while the other eye will undergo phacoemulsification with Trypan Blue capsule staining (study eye). Both eyes will undergo intraocular lens implantation. Preoperative and four-week postoperative quantitative and qualitative morphometric endothelial cell analyses of the cornea will be performed using noncontact specular microscopy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with bilateral cataract and diabetic retinopathy

Exclusion Criteria:

* History of ocular surgery Active
* ocular inflammation Corneal opacities
* Pseudoexfoliation syndrome
* Anterior chamber flare and (or) other signs of possibly altered blood - queous barrier
* Iris neovascularization (rubeosis)
* Uncontrolled glaucoma
* Congenital or traumatic cataracts
* History or present chronic use of topical or systemic steroids
* Poor papillary dilatation (<6 mm)
* Specular microscopy cell density < 2000 cell/mm2
* Patients who experienced complications fromphacoemulsification

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-07-25 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Endothelial cell density | 4 weeks

SECONDARY OUTCOMES:
Endothelial cell coefficient of variation | 4 weeks
Percent of hexagonal cells | 4 weeks
Mean corneal thickness | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abdelmotaal H, Abdelazeem K, Hussein MS, Omar AF, Ibrahim W. Safety of Trypan Blue Capsule Staining to Corneal Endothelium in Patients with Diabetic Retinopathy. J Ophthalmol. 2019 Mar 27;2019:4018739. doi: 10.1155/2019/4018739. eCollection 2019. PMID 31032113